## ENHANCING ENGAGEMENT WITH DIGITAL MENTAL HEALTH CARE STUDY00010958

11/14/2023

NCT04507360

## University of Washington Consent Form

This page gives you information to help you decide whether or not to be in this research study. Being in the study is voluntary. Please read this carefully. After doing so, you can decide whether or not you want to be in the study.

**Purpose:** The purpose of the study is to better understand how self-help mental health resources can help people overcome negative thinking and support healthier thought processes. This study is being conducted by researchers at the University of Washington in partnership with Mental Health America.

**Procedure:** We will be testing three different mental health resources to see how well each method works. Participants are each randomly assigned, like flipping a coin, to work with one of those resources for four weeks. You will be notified of your randomly assigned condition via email after agreeing to participate in the study. Each week, you will be asked to fill out a survey about your thinking patterns and mental well-being. These surveys will be sent to you via SMS text message or email, and we think they will each take less than 10 minutes to complete. You will be given a self-guided mental health resource to be used up to three times a week for less than 5 minutes each time.

Compensation: You may earn between up to \$40-60 for your participation in the study. After agreeing to participate in the study, you will be randomized to a mental health resource condition. Incentive amounts earned will be tied to effort demonstrated in completing requested tasks, and you will receive more specific information regarding incentives after randomization. Incentives will be sent via email from mentalhealthstudy@uw.edu in the form of Amazon gift codes.

**Benefits:** There will be no direct benefit to you from participating in this study. However, through the resources in this study, you may learn about how to manage negative thinking.

**Risks:** Thinking about and sharing information on your mental health and well-being may make you feel upset. The resources were designed to avoid harmful content generation, but there is a possibility that the content might be upsetting to you. Also, our surveys ask for information that may be sensitive and could make you feel uncomfortable (e.g., "Over the last two weeks, how often did you feel down, depressed, or hopeless"). Neither responses to survey questions nor the resources will be actively monitored by a human and should not be used as a "cry for help" outlet. If you are experiencing emotional distress and/or thoughts of self-harm or suicide, text MHA to 741741 or call or text 988.

There are no costs to you for participating in the study. However, taking surveys or using the resources with your mobile phone may count against your mobile data plan. You may change your settings to only use Wi-Fi connections to manage how this data collection will affect your plan. Alternatively, you may take the surveys and use the resources with a computer.

**Data Collection and Sharing:** All the information you provide will be confidential. We will collect your name, email address, and cell phone number, but that information will be stored separately from other study data. Resource usage data will be de-identified to the best of our extent and will not be shared

outside our research groups at Mental Health America and the University of Washington. The data will be analyzed to assess the resources. It is possible that the information we obtain from you for this study might be used for future studies. If we remove anything that might identify you, that information may then be used for future research studies or given to another investigator without getting additional permission from you. If we want to use or share study information that might identify you, a review board will decide whether we need to get additional permission from you.

**Participation:** Participation in this study is completely voluntary. You can refuse participation or stop participating at any time without penalty or loss of benefits to which you are otherwise entitled.

**Study Funding:** This study is funded by the National Institute of Mental Health (NIMH). We have a Certificate of Confidentiality from NIMH which allows us to keep your identifiable research information confidential from legal proceedings or in response to a legal request unless you give us permission to release it. You or a member of your family can share information about yourself or your part in this research if you wish. There are some limits to this protection, including reporting things like child or elder abuse, monitoring by the agencies conducting the research, and others as listed elsewhere in this consent form. The Certificate expires when the NIMH funding for this study ends. Currently this date is November 30, 2024. Data collected prior to expiration will continue to be protected.

Contact Us: We are here to help you understand the study. Please ask us any questions you may have, even about things that are not in this document. Please contact us at mentalhealthstudy@uw.edu with any questions about the study or your participation in the study. If you think you have been harmed from being in the study, please email the principal investigators Mike Pullmann (pullmann@uw.edu) and Tim Althoff (althoff@cs.washington.edu). If you have questions about your rights as a research participant, you can call the University of Washington Human Subjects Division at (206) 543-0098 or hsdinfo@uw.edu.

By ticking this box, you are agreeing to participate in this study. You are also confirming that you are at least 18 years old. Be sure that questions about the study have been answered and that you understand what you are being asked to do. You may contact us if you think of a question later. You are free to stop participating in the study at any time. To save a copy of this consent form, you can use this link.